CLINICAL TRIAL: NCT03454542
Title: Assessment of Comfort and Ocular Surface Parameters With Novel Designs of Daily Disposable Silicone Hydrogel Contact Lenses (BASS)
Brief Title: Assessment of Comfort & Ocular Surface Parameters w Novel Designs of Daily Disposable Silicone Hydrogel Contact Lenses
Acronym: BASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P/626/17/M
Record Dates: First submitted 2018-02-20; First posted 2018-03-06 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-03

CONDITIONS: Visual Acuity; Contact Lens Comfort

STUDY DESIGN:
Intervention Model Description: This will be a double-masked, cross-over, bilateral wear study design with five (5) study visits across three (3) study visit days. Participants will be dispensed and wear both the initial and modified lens design for a total of six (6) hours each on two (2) separate visit days, with the order of lens wear being randomized; participants will be allowed to leave the CCLR on their lens wearing days between dispense and follow-up visit.
Who Masked: Participant, Investigator
Masking Description: This will be a double-masked study, with both the study participants and study investigators being masked to the order of lens wear for the initial and modified DD lens design. Study lenses will be dispensed to the participants at V2 and V4 by unmasked research assistants from paper cups. Lenses and blister-pack solution will be directly transferred into the paper cups, and only the paper cups will be taken to the examination room where lenses are being dispensed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menicon DSRB Redesign (Experimental): Menicon DSRB Modified Lens Design is a single use contact lens with revised thickness specifications worn for 6 hours or more.
  Interventions: Device: Menicon Modified Lens Design
- Menicon DSRB Original Design (Active Comparator): Menicon DSRB Initial Lens Design is a single use contact lens with the original thickness specifications worn for 6 hours or more.
  Interventions: Device: Menicon Modified Lens Design

INTERVENTIONS:
Device: Menicon Modified Lens Design — Randomized in a daily wear, single day (6 hours or more) evaluation

SUMMARY:
A comparison of two lens designs manufactured in the same material. The hypothesis is the subjectively rated performance of comfort, vision and lens handling will be better with the modified design compared to the initial design

DETAILED DESCRIPTION:
The objectives of the study are

1. to identify possible reasons for the different comfort and vision experience in Japanese CL wearers compared to Caucasian CL wearers and
2. to assess whether the modification of lens thickness in the optical zone results in increased comfort and reduced visual acuity fluctuations in Caucasian eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is of Caucasian heritage;
5. Habitually wears soft spherical daily disposable contact lenses with a power between

   -0.50 to -2.75D (inclusive);
6. Demonstrates an acceptable fit with both study CL designs (initial & modified);
7. Is correctable to a visual acuity of 0.20 LogMAR (approximately 20/30) or better (in each eye) with both study CL designs;
8. Has a manifest cylindrical spectacle refraction that does not exceed -1.00DC in either eye;
9. Should own a wearable pair of spectacles. -

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by self-report);
7. Is aphakic;
8. Has undergone refractive error surgery; -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Participant's subjective rating of comfort, Questionnaire | 2 Days
  Participants rate their eye comfort by subjective questionnaire (non-annotated scale, 0-100, 0=painful, 100=can't feel the lenses)
Participant's subjective rating of vision, Questionnaire | 2 Days
  Participants rate their vision by subjective questionnaire (non-annotated scale, 0-100, 0=not at all sharp/clear, 100=sharp/clear
Participant's subjective rating of lens handling, Questionnaire | 2 Days
  Participants rate their ability to handle the contact lens by subjective questionnaire (non-annotated scale, 0-100, 0=very difficult, 100=very easy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada